CLINICAL TRIAL: NCT02996812
Title: Subcutaneous Injection of Exendin (9-39) in Subjects With Hyperinsulinemic Hypoglycemia Post-Bariatric Surgery
Brief Title: Evaluation of Single Ascending Doses of Subcutaneous Exendin 9-39 in Patients With Post-Bariatric Hypoglycemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tracey McLaughlin (Other)
Responsible Party: Sponsor-Investigator, Tracey McLaughlin, Associate Professor of Medicine (Endocrinology), Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 34054
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Hyperinsulinemia Hypoglycemia
Keywords: Post-bariatric hypoglycemia; Non-insulinoma pancreatogenous hypoglycemia syndrome; Late dumping syndrome
MeSH Terms: conditions — Congenital Hyperinsulinism | interventions — exendin (9-39)

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose A (Active Comparator): Subcutaneous injection of Dose A of Exendin (9-39)
  Interventions: Drug: Exendin (9-39)
- Dose B (Active Comparator): Subcutaneous injection of Dose B of Exendin (9-39)
  Interventions: Drug: Exendin (9-39)
- Dose C (Active Comparator): Subcutaneous injection of Dose C of Exendin (9-39)
  Interventions: Drug: Exendin (9-39)
- Dose D (Active Comparator): Subcutaneous injection of Dose D of Exendin (9-39)
  Interventions: Drug: Exendin (9-39)

INTERVENTIONS:
Drug: Exendin (9-39)

SUMMARY:
This study is designed to evaluate the safety, efficacy, and pharmacokinetic profile of single ascending doses of exendin 9-39 administered by subcutaneous route in subjects with post-bariatric hypoglycemia.

DETAILED DESCRIPTION:
Post-Bariatric Hypoglycemia (PBH) is a debilitating rare disease afflicting 0.2-6.9% of post-bariatric patients, characterized by repeated severe hypoglycemic episodes with neuroglycopenic symptoms and marked disability. There are no effective medical therapies.

While the cause is not known, exaggerated postprandial secretion of glucagon-like peptide-1 (GLP-1) as a result of altered nutrient transit likely plays a major role. GLP-1 is an incretin hormone secreted primarily by the distal ileum that contributes to postprandial glucose regulation. Exendin 9-39 (Ex9) is a specific GLP-1 receptor antagonist, that when given via continuous IV infusion, has been shown to effectively prevent postprandial hypoglycemia in patients with PBH. Subcutaneous (SC) injection of Ex9 may represent a safe, effective and practical therapeutic approach to treating PBH.

ELIGIBILITY:
Inclusion Criteria:

* Post-bariatric surgery more than 6 months prior to signing the informed consent
* Reported history of Whipple's triad: the occurrence of hypoglycemic symptoms associated with blood glucose of ≤55 mg/dL, and resolution with glucose or carbohydrate administration.
* Symptomatic hypoglycemia during the baseline/screening OGTT, as defined by the presence of plasma glucose ≤55 mg/dL with concomitant autonomic and/or neuroglycopenic symptoms.

Exclusion Criteria:

* Patients currently using sulfonylureas or other medications that may interfere with glucose metabolism within 5 half-lives of drug.
* Participation in any clinical investigation within 4 weeks prior to dosing
* History of or current insulinoma
* Active infection or significant acute illness within 2 weeks prior to dosing
* Female patients who are pregnant or lactating
* Women of childbearing potential and not utilizing effective contraceptive methods
* Inadequate end organ function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Treatment effect on plasma glucose | 0-180 minutes following initiation of oral glucose tolerance test (OGTT) conducted after treatment.
  Magnitude of plasma glucose nadir during repeat OGTT after treatment

SECONDARY OUTCOMES:
Treatment effect on symptoms of hypoglycemia | 0-180 minutes following initiation of OGTT
  Response rate in symptom score during repeat OGTT after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Tracey McLaughlin, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No